CLINICAL TRIAL: NCT02993107
Title: Peanut Allergy Oral Immunotherapy Study of AR101 for Desensitization in Children and Adults (PALISADE) Follow-on Study
Brief Title: PALISADE Follow-on Study (ARC004)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC004
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Peanut Allergy
Keywords: AR101; Characterized Peanut Allergen; CPNA (Characterized Peanut Allergen); OIT (oral immunotherapy); Peanut Allergy; Allergy; Peanut-Allergic Children; Peanut-Allergic Adults; Desensitization; PALISADE
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Crossovers) (Other): Subjects who complete the placebo arm of ARC003 and consent to enroll in ARC004 (Group-1) will cross over to active treatment with AR101 using the same dosing regimen used in ARC003 in open-label fashion. Group 1 subjects may also be assigned to cohorts which test the gradual lengthening of dosing intervals. Following the completion of their longest tested dosing interval, Group 1 subjects will undergo an exit double-blinded placebo-controlled food challenge (DBPCFC).
  Interventions: Biological: AR101
- Group 2 (Active Rollovers) (Other): Subjects who successfully complete the active arm of ARC003 and consent to enroll in ARC004 (Group-2) will consecutively enter treatment with AR101 in one of three cohorts which will test alternate dosing intervals. There will be a DBPCFC at the completion of the subject's longest tested dosing interval.
  Interventions: Biological: AR101

INTERVENTIONS:
Biological: AR101 — AR101 powder provided in capsules & sachets

SUMMARY:
The purpose of this study is to demonstrate the safety, tolerability, and efficacy of AR101 through oral immunotherapy (OIT) in peanut-allergic children and adults who have completed the ARC003 study.

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, 2-arm follow-on study of the safety, tolerability, and efficacy of AR101 in peanut-allergic individuals who have completed the ARC003 study. This study will explore alternative dosing regimens during extended maintenance with AR101.

ELIGIBILITY:
Key Inclusion Criteria:

* Completion of the ARC003 study
* Written informed consent and/or assent from subjects/guardians as appropriate
* Use of effective birth control by sexually active female subjects of child-bearing potential

Key Exclusion Criteria:

* Early discontinuation from the ARC003 study
* Meets any longitudinally applicable ARC003 study exclusion criteria
* (Group 2 only) Failure to tolerate ≥ 443 mg cumulative of peanut protein with no or mild symptoms in the ARC003 study Exit DBPCFC
* Any other condition that, in the opinion of the Investigator, precludes participation for reasons of safety

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 388 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Director — Aimmune Regulatory Affairs
Locations (64):
- United States (47):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Sean N. Parker Center for Allergy Research at Stanford University Packard-El Camino Hospital, Mountain View, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, APC, San Diego, California
  - Rady Children's Hospital, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado Allergy & Asthma Centers, P.C., Centennial, Colorado
  - National Jewish Health, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Sarasota Clinical Research, Sarasota, Florida
  - University of South Florida Asthma, Allergy, and Immunology Clinical Research Unit, Tampa, Florida
  - Atlanta Allergy & Asthma Clinic, PA, Marietta, Georgia
  - Idaho Allergy and Research, dba Idaho Research, Eagle, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - IU North Riley Children's Specialist, Carmel, Indiana
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Div. of Allergy & Immunology, Boston, Massachusetts
  - Michigan Medicine, Michigan Clinical Research Unit, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Plymouth, Minnesota
  - Children's Mercy on Broadway, Kansas City, Missouri
  - Nebraska Medical Research Institute Inc., Bellevue, Nebraska
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Icahn School of Medicine at Mount Sinai, Clinical Research Unit, New York, New York
  - University of North Carolina at Chapel Hill, Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baker Allergy, Asthma & Dermatology, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research, LLC, Charleston, South Carolina
  - Le Bonheur Children's Hospital - Outpatient Building, Memphis, Tennessee
  - 'Specially for Children Allergy, Asthma and Immunology Clinic, Austin, Texas
  - Children's Health, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Benaroya Research Inst. at Virginia Mason; Virginia Mason Medical Center, Seattle, Washington
  - Asthma Inc Clinical Research Center, Seattle, Washington
- Canada (5):
  - Triple A Lab, Hamilton, Ontario
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Inc., Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Germany (2):
  - Charité Universitaetsmedizin Berlin, Berlin
  - University of Frankfurt, Frankfurt am Main
- Cork University Hospital, Cork, Ireland
- Azienda Ospedaliera di Padova, Padua, Italy
- Netherlands (2):
  - Beatrix Children's Hospital, University Medical Center Groningen, Groningen
  - University Medical Center Groningen, Groningen
- Spain (3):
  - Hospital Gregorio Marañón, Madrid
  - H. Infantil Universitario Niño Jesús, Madrid
  - Hospital Clinico San Carlos, Madrid
- Sachsska Children and Youth Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Guy & St Thomas' NHS foundation Trust, London
  - Central Manchester University Hospitals, NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blumchen K, Kleinheinz A, Klimek L, Beyer K, Anagnostou A, Vogelberg C, Butovas S, Ryan R, Norval D, Zeitler S, Du Toit G. Post hoc analysis examining symptom severity reduction and symptom absence during food challenges in individuals who underwent oral immunotherapy for peanut allergy: results from three trials. Allergy Asthma Clin Immunol. 2023 Mar 13;19(1):21. doi: 10.1186/s13223-023-00757-8. PMID 36915184
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Placebo Crossovers): Received AR101 during IDE (day 1, 0.5 to 3 or 6 mg; day 2, 3 mg), up-dosing (3-300 mg/day for 22-40 weeks, with dose escalations every 2 weeks), and maintenance (300 mg/day for 24-28 weeks).
- Group 2: Cohort 1 (Active Rollovers): Received 300 mg/day (once daily, QD) peanut protein for 28 weeks
- Group 2: Cohort 2 (Active Rollovers): Received 300 mg peanut protein every other day (QOD) for 4 weeks, then twice weekly (BIW) for 24 weeks for a total of 28 weeks
- Group 2: Cohort 3A (Active Rollovers): Received 300 mg/day peanut protein for 56 weeks
- Group 2: Cohort 3B (Active Rollovers): Received 300 mg/day peanut protein for 28 weeks, QOD for 4 weeks, then BIW for 24 weeks (total of 56 weeks)
- Group 2: Cohort 3C (Active Rollovers): Received 300 mg/day peanut protein for 28 weeks, QOD for 4 weeks, BIW for 24 weeks, then once weekly (QW) for 28 weeks (total of 84 weeks)
Period: Overall Study
Arm/Group | Group 1 (Placebo Crossovers) | Group 2: Cohort 1 (Active Rollovers) | Group 2: Cohort 2 (Active Rollovers) | Group 2: Cohort 3A (Active Rollovers) | Group 2: Cohort 3B (Active Rollovers) | Group 2: Cohort 3C (Active Rollovers)
Started | 113 | 120 | 50 | 35 | 34 | 36
Adverse Event | 12 | 4 | 1 | 1 | 3 | 5
Physician Decision | 1 | 0 | 1 | 0 | 0 | 0
Withdrawal by Subject | 32 | 7 | 7 | 3 | 6 | 2
Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1
Sponsor Decision | 4 | 0 | 1 | 1 | 0 | 4
Protocol Deviation | 0 | 0 | 0 | 0 | 1 | 0
Other Reasons | 2 | 1 | 1 | 1 | 2 | 3
Completed | 62 | 107 | 39 | 29 | 22 | 21
Not Completed | 51 | 13 | 11 | 6 | 12 | 15

BASELINE CHARACTERISTICS:
Population: A total of 388 subjects were enrolled. However, only 381 received any amount of treatment and were included in the Safety population, which includes all subjects who received at least one dose of open-label study treatment in any cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Placebo Crossovers) | Group 2: Cohort 1 (Active Rollovers) | Group 2: Cohort 2 (Active Rollovers) | Group 2: Cohort 3A (Active Rollovers) | Group 2: Cohort 3B (Active Rollovers) | Group 2: Cohort 3C (Active Rollovers) | Total
Number analyzed (Participants) | 111 | 117 | 48 | 35 | 34 | 36 | 381
Age, Customized [Count of Participants; unit: Participants]
  Age 18-55 years | 11 | 8 | 2 | 4 | 3 | 2 | 30
  Age 4-17 years | 100 | 109 | 46 | 31 | 31 | 34 | 351
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 55 | 22 | 16 | 13 | 17 | 162
  Male | 72 | 62 | 26 | 19 | 21 | 19 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 3 | 4 | 1 | 1 | 31
  Not Hispanic or Latino | 98 | 108 | 45 | 31 | 33 | 35 | 350
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 7 | 14 | 7 | 3 | 1 | 3 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 3 | 1 | 0 | 0 | 0 | 7
  White | 86 | 92 | 33 | 28 | 30 | 28 | 297
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 8 | 7 | 4 | 2 | 4 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Ages 4-17 With Treatment-related Adverse Events (TEAE)
Description: Percentage of subjects ages 4-17 with at-least 1 TEAE, including serious adverse events, during the overall study period. The percentage of subjects reporting at least 1 TEAE by maximum reported severity is also presented using the 5-point CTCAE severity grading scale. All safety evaluations were conducted using the safety population (all subjects who received at least 1 dose of AR101 during ARC004), age 4-17 years. Safety data are presented for group 1 (former placebo) and Group 2 data are divided into columns for cohort 1 (QD), cohort 2 (overall), cohort 3A (QD), and cohorts 3B and 3C (overall).
Time Frame: Up to 126 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 (Overall): Received AR101 during IDE (day 1, 0.5 to 3 or 6 mg; day 2, 3 mg), up-dosing (3-300 mg/day for 22-40 weeks, with dose escalations every 2 weeks), and maintenance (300 mg/day for 24-28 weeks).
- Group 2: Cohort 1 (QD): Received 300 mg/day (once daily, QD) peanut protein for 28 weeks
- Group 2: Cohort 2 (Overall): Received 300 mg peanut protein every other day (QOD) for 4 weeks, then twice weekly (BIW) for 24 weeks for a total of 28 weeks
- Group 2: Cohort 3A (QD): Received 300 mg/day peanut protein for 56 weeks
- Group 2: Cohort 3B (Overall): Cohort 3B: Received 300 mg/day peanut protein for 28 weeks, QOD for 4 weeks, then BIW for 24 weeks (total of 56 weeks)
- Group 2: Cohort 3C (Overall): Cohort 3C: Received 300 mg/day peanut protein for 28 weeks, QOD for 4 weeks, BIW for 24 weekly (QW) for 28 weeks (total 84 weeks)
Arm/Group | Group 1 (Overall) | Group 2: Cohort 1 (QD) | Group 2: Cohort 2 (Overall) | Group 2: Cohort 3A (QD) | Group 2: Cohort 3B (Overall) | Group 2: Cohort 3C (Overall)
Number analyzed (Participants) | 100 | 109 | 46 | 31 | 31 | 34
Participants
  All AEs | 98 | 90 | 36 | 27 | 28 | 33
  SAEs | 0 | 1 | 0 | 0 | 1 | 1
  Grade 1: Mild | 37 | 58 | 22 | 15 | 13 | 12
  Grade 2: Moderate | 58 | 29 | 14 | 12 | 15 | 18
  Grade 3: Severe | 3 | 3 | 0 | 0 | 0 | 3
  Grade 4: Life-Threatening | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5: Death | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Subjects Ages 4-17 Responding to Each Challenge Dose at Exit DBPCFC (Double-blind, Placebo-controlled Food Challenge)
Description: The percentage of subjects who tolerated each the of 300 mg, 600 mg, 1000 mg, or 2000 mg challenge doses with no more than mild symptoms at exit DBPCFC. Analyses based on DBPCFCs used the completer population (age 4-17 years).
Time Frame: Up to 126 weeks
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Group 1 (Placebo Crossovers): Received AR101 during IDE (day 1, 0.5 to 3 or 6 mg; day 2, 3 mg), up-dosing (3-300 mg/day for 22-40 weeks, with dose escalations every 2 weeks), and maintenance (300 mg/day for 24-28 weeks) (age 4-17).
Arm/Group | Group 1 (Placebo Crossovers) | Group 2: Cohort 1 (Active Rollovers) | Group 2: Cohort 2 (Active Rollovers) | Group 2: Cohort 3A (Active Rollovers) | Group 2: Cohort 3B (Active Rollovers) | Group 2: Cohort 3C (Active Rollovers)
Number analyzed (Participants) | 72 | 103 | 38 | 26 | 22 | 21
Percent of participants
  Percentage (and 95% CI) tolerating 300 mg | 98.6 [92.5 to 100] | 98.1 [93.2 to 99.8] | 94.7 [82.3 to 99.4] | 100.0 [86.8 to 100.0] | 81.8 [59.7 to 94.8] | 90.5 [69.6 to 98.8]
  Percentage (and 95% CI) tolerating 600 mg | 86.1 [75.9 to 93.1] | 89.3 [81.7 to 94.5] | 71.1 [54.1 to 84.6] | 96.2 [80.4 to 99.9] | 77.3 [54.6 to 92.2] | 76.2 [52.8 to 91.8]
  Percentage (and 95% CI) tolerating 1000 mg | 72.2 [60.4 to 82.1] | 80.6 [71.6 to 87.7] | 57.9 [40.8 to 73.7] | 96.2 [80.4 to 99.99] | 68.2 [45.1 to 86.1] | 66.7 [43.0 to 85.4]
  Percentage (and 95% CI) tolerating 2000 mg | 51.4 [39.3 to 63.3] | 48.5 [38.6 to 58.6] | 36.8 [21.8 to 54.0] | 80.8 [60.6 to 93.4] | 45.5 [24.4 to 67.8] | 42.9 [21.8 to 66.0]

ADVERSE EVENTS:
Time Frame: 28 months
Description: The data is presented separately for the 4-17 year old age group (children and adolescents) and 18-55 year old age group (adults).
Groups:
- Group 1 (Age 4-17 Overall); Group 1 (Age 18-55 Overall): Received AR101 during IDE (day 1, 0.5 to 3 or 6 mg; day 2, 3 mg), up-dosing (3-300 mg/day for 22-40 weeks, with dose escalations every 2 weeks), and maintenance (300 mg/day for 24-28 weeks).
- Group 2: Cohort 1 (Age 4-17 QD); Group 2: Cohort 1 (Age 18-55 QD): Received 300 mg/day (once daily, QD) peanut protein for 28 weeks.
- Group 2: Cohort 2 (Age 4-17 Overall); Group 2: Cohort 2 (Age 18-55 Overall): Received 300 mg peanut protein every other day (QOD) for 4 weeks, then twice weekly (BIW) for 24 weeks for a total of 28 weeks.
- Group 2: Cohort 3A (Age 4-17 QD); Group 2: Cohort 3A (Age 18-55 QD): Received 300 mg/day peanut protein for 56 weeks.
- Group 2: Cohort 3B (Age 4-17 Overall); Group 2: Cohort 3B (Age 18-55 Overall): Cohort 3B: Received 300 mg/day peanut protein for 28 weeks, QOD for 4 weeks, then BIW for 24 weeks (total of 56 weeks).
- Group 2: Cohort 3C (Age 4-17 Overall); Group 2: Cohort 3C (Age 18-55 Overall): Cohort 3C: Received 300 mg/day peanut protein for 28 weeks, QOD for 4 weeks, BIW for 24 weekly (QW) for 28 weeks (total 84 weeks).
Arm/Group | Group 1 (Age 4-17 Overall) | Group 2: Cohort 1 (Age 4-17 QD) | Group 2: Cohort 2 (Age 4-17 Overall) | Group 2: Cohort 3A (Age 4-17 QD) | Group 2: Cohort 3B (Age 4-17 Overall) | Group 2: Cohort 3C (Age 4-17 Overall) | Group 1 (Age 18-55 Overall) | Group 2: Cohort 1 (Age 18-55 QD) | Group 2: Cohort 2 (Age 18-55 Overall) | Group 2: Cohort 3A (Age 18-55 QD) | Group 2: Cohort 3B (Age 18-55 Overall) | Group 2: Cohort 3C (Age 18-55 Overall)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/109 | 0/46 | 0/31 | 0/31 | 0/34 | 0/11 | 0/8 | 0/2 | 0/4 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/109 | 0/46 | 0/31 | 1/31 | 1/34 | 0/11 | 1/8 | 0/2 | 0/4 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 98/100 | 90/109 | 36/46 | 27/31 | 28/31 | 33/34 | 10/11 | 6/8 | 1/2 | 2/4 | 2/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Age 4-17 Overall) (N=100) | Group 2: Cohort 1 (Age 4-17 QD) (N=109) | Group 2: Cohort 2 (Age 4-17 Overall) (N=46) | Group 2: Cohort 3A (Age 4-17 QD) (N=31) | Group 2: Cohort 3B (Age 4-17 Overall) (N=31) | Group 2: Cohort 3C (Age 4-17 Overall) (N=34) | Group 1 (Age 18-55 Overall) (N=11) | Group 2: Cohort 1 (Age 18-55 QD) (N=8) | Group 2: Cohort 2 (Age 18-55 Overall) (N=2) | Group 2: Cohort 3A (Age 18-55 QD) (N=4) | Group 2: Cohort 3B (Age 18-55 Overall) (N=3) | Group 2: Cohort 3C (Age 18-55 Overall) (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Age 4-17 Overall) (N=100) | Group 2: Cohort 1 (Age 4-17 QD) (N=109) | Group 2: Cohort 2 (Age 4-17 Overall) (N=46) | Group 2: Cohort 3A (Age 4-17 QD) (N=31) | Group 2: Cohort 3B (Age 4-17 Overall) (N=31) | Group 2: Cohort 3C (Age 4-17 Overall) (N=34) | Group 1 (Age 18-55 Overall) (N=11) | Group 2: Cohort 1 (Age 18-55 QD) (N=8) | Group 2: Cohort 2 (Age 18-55 Overall) (N=2) | Group 2: Cohort 3A (Age 18-55 QD) (N=4) | Group 2: Cohort 3B (Age 18-55 Overall) (N=3) | Group 2: Cohort 3C (Age 18-55 Overall) (N=2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 2 | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 8 | 5 | 4 | 1 | 3 | 6 | 2 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 17 | 6 | 5 | 0 | 2 | 3 | 3 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 38 | 11 | 7 | 5 | 7 | 16 | 5 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 31 | 9 | 6 | 5 | 6 | 4 | 6 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 1 | 4 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip pruritus (Gastrointestinal disorders) | 11 | 3 | 2 | 2 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 8 | 3 | 4 | 3 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 33 | 9 | 9 | 5 | 5 | 5 | 6 | 0 | 1 | 1 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pruritus (Gastrointestinal disorders) | 17 | 6 | 5 | 4 | 3 | 7 | 3 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 6 | 0 | 2 | 2 | 2 | 4 | 3 | 0 | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue pruritus (Gastrointestinal disorders) | 11 | 3 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 5 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 42 | 18 | 6 | 6 | 9 | 9 | 3 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 9 | 3 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 9 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 6 | 0 | 2 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 24 | 20 | 4 | 8 | 6 | 13 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 17 | 7 | 0 | 5 | 2 | 10 | 4 | 1 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 6 | 1 | 1 | 5 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 8 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 4 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 2 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 9 | 7 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 7 | 7 | 1 | 1 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 16 | 5 | 5 | 5 | 5 | 9 | 3 | 0 | 0 | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 4 | 5 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 6 | 1 | 0 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 2 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 23 | 20 | 6 | 3 | 5 | 7 | 5 | 4 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 10 | 9 | 1 | 5 | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 4 | 5 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary physical examination abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eating disorder symptom (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 27 | 12 | 12 | 8 | 5 | 14 | 1 | 1 | 0 | 1 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 0 | 4 | 6 | 2 | 0 | 1 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 16 | 8 | 8 | 10 | 16 | 3 | 1 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 1 | 3 | 5 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 8 | 6 | 2 | 4 | 6 | 1 | 0 | 0 | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 7 | 4 | 7 | 6 | 8 | 3 | 0 | 0 | 2 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 28 | 7 | 2 | 3 | 4 | 7 | 6 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 18 | 8 | 4 | 3 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 32 | 15 | 9 | 5 | 5 | 9 | 7 | 0 | 0 | 0 | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 17 | 3 | 2 | 2 | 2 | 7 | 2 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 7 | 2 | 1 | 2 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 7 | 6 | 1 | 7 | 5 | 4 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 14 | 6 | 1 | 1 | 3 | 5 | 1 | 1 | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 37 | 16 | 6 | 7 | 6 | 9 | 1 | 0 | 1 | 2 | 0 | 0
Rhinoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sclerotherapy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 6 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02993107/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT02993107/SAP_001.pdf